CLINICAL TRIAL: NCT00221767
Title: Prospective Comparative Multicenter Study on the Medico-economical Impact of the Brindley Technique in the Management of Neurogenic Bladder in Patients With Injured Spinal Cord
Brief Title: Medico-economical Impact of the Brindley Neurosurgical Technique in France
Acronym: BRINDLEY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 9415-04; 2004-001
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Spinal Cord Injuries; Neurogenic Bladder Disorder; Paraplegia; Quadriplegia
Keywords: Neurogenic bladder; electric stimulation therapy; urinary tract infection; urinary incontinence; spinal cord injuries; spinal nerve roots; nonRandomized Controlled Trials; open Study
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic; Paraplegia; Quadriplegia; Urinary Tract Infections; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Brindley technique (bladder system)
  Interventions: Device: Brindley technique (bladder system)
- 2 (No Intervention): Reference group

INTERVENTIONS:
Device: Brindley technique (bladder system) — Sacral posterior rhizotomies and implantation of Brindley device on sacral anterior roots
  Arms: 1

SUMMARY:
Bladder dysfunction is a major problem in patients with complete spinal cord lesions. For patients presenting incontinence or risk for kidney, two major conventional alternatives are possible : conservative therapies (muscarinic receptor antagonists, vanilloids drugs and botulinum toxin in association with catheterization) and surgical techniques intervening in the nervous and urinary system.

Among these last alternatives, the Brindley technique (anterior sacral root stimulation with posterior rhizotomy) is the only technique allowing for the restauration of bladder function, continence, and micturition. The purpose of the study is to compare the Brindley technique with the first conventional approach in France from a medical and economical point of view.

DETAILED DESCRIPTION:
Background : In paraplegic and tetraplegic patients with suprasacral lesion, bladder overactivity leads to incontinence and is frequently associated with detrusor-sphincter dyssynergia which is responsible for residual postvoiding (high infectious risk) and intravesical high pressure (risk for kidney). The Brindley technique allows to restore a voluntary voiding of the bladder and an effective continence. Electrodes are fixed to anterior sacral roots in order to obtain micturition. Posterior sacral root rhizotomy suppress detrusor and sphincter overactivity, improves continence and thus protects bladder and kidney (low pressure bladder filling). Currently in France, 100 new patients could benefit from this innovative technique among the 1000 patients with spinal cord injury

Objective :To compare the cost/effectiveness ratio of the Brindley technique approach to that of the reference group (muscarinic receptor antagonists + catheterization or reflex micturition)at one year, in patient with neurogenic bladder.

In this prospective, comparative, non-randomized, multicenter study, the eligible patients are included according to the following ratio : 2:1 (Brindley : Reference ). The complete suprasacral spinal cord injured patients with an overactive neurogenic bladder, incontinence and/or risk of kidney/bladder injury) are the population studied. The spinal cord injury must be clinically stable for at least 3 months.

primary outcome :Proportion of patients showing a complete voluntary (including electrostimulation) micturition after one year.

Secondary outcome : Bladder capacity (cystometry), costs, incidence of urinary infections, incontinence, autonomic hyperreflexia (AHR), defecation, quality of life, lower limbs spasticity.

Patient follow-up :Visits must be planned at 1, 3, 6, 9 and 12 months: A classical clinical exam and a specific exam (evaluation of AHR, Ashworth and Penn Score) at 6 and 12 months and the following complementary exams at 3, 6 and 12 months: urodynamic testing and intravenous urography, retrograde ureterocystography and bladder echography at 12 months.

Population size : A total number of 99 patients must be enrolled to achieve the fixed goals (66 patients in the Brindley group and 33 patients in the Reference group).

ELIGIBILITY:
Inclusion Criteria:

* Patient with a complete suprasacral spinal cord injury proved by a clinical exam (perineal reflex preserved) and MRI.
* Clinically stable spinal cord injury for at least 6 months (verified by MRI)
* Patient with an overactive neurogenic bladder (urodynamic testing), incontinence (specific patient diary) and/or risk for the bladder/kidney (intravenous urography, cystography)
* signed informed consent

Exclusion Criteria:

* Injured sacral medullar centers or injured sacral roots
* Non contractile bladder
* Pregnancy or breast feeding
* Contraindication linked to neurostimulator implantation: unwounded cutaneous lesion, prolonged septic state, blood coagulation deficiency, known allergy to one component of the implanted medical device (silicone, platinum, iridium)
* Incapacity to receive an informed consent, incapacity to follow all the study schedule,
* patient not protected by social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2005-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients showing a complete voluntary (including electrostimulation) micturition | At 3 months, 6 months and at one year

SECONDARY OUTCOMES:
Bladder capacity (cystometry) | At 3 months, 6 months and after one year
costs | At 3 months, 6 months, 9 months and at one year
incidence of urinary infections | At visit 3, 6 and at one year
incontinence | At 3 months, 6 months and at one year
autonomic hyperreflexia (AHR) | At 3 months, 6 months, and at one year
defecation | at 3 months, 6 months and at one year
quality of life | at 6 months and at one year
lower limbs spasticity | at 3 months, 6 months and at one year

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Rodolphe Vignes, Doctor, Principal Investigator — University Hospital, Bordeaux; Geneviève Chêne, Professor, Study Chair — University Hospital, Bordeaux
Locations (1):
- Neurochirurgie A - Hôpital Pellegrin , Place Amélie Raba-Léon, Bordeaux, France